CLINICAL TRIAL: NCT02734186
Title: Effect of Concomitant Mansonella Perstans Microfilaremia on Immune Responses Following Single Dose Praziquantel in Subjects With Schistosomiasis: A Pilot Study
Brief Title: Effect of Concomitant Mansonella Perstans Microfilaremia on Immune Responses Following Single Dose Praziquantel in People With Schistosomiasis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 999916084; 16-I-N084
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-12-14

CONDITIONS: Schistosomiasis
Keywords: Filariasis; Schistosoma Mansoni; Coinfection
MeSH Terms: conditions — Schistosomiasis; Filariasis; Coinfection | interventions — Praziquantel

ARMS (2):
- Sh (Experimental): Mono infected with Schistosoma haematobium
  Interventions: Drug: Praziquantel
- ShMp (Experimental): Coinfected with Schistosoma haematobium andMansonella perstans
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Praziquantel — Anthelminthic

SUMMARY:
Background:

Schistosomiasis is a chronic infection. It is caused by parasitic worms called Schistosoma haematobium (Sh) that are spread by snails that live in rivers. It can lead to liver problems or bladder cancer. Praziquantel (PZQ) is a drug used to treat this infection. After taking it, some people develop increased resistance to reinfection with Sh. Some people with Sh infection can be infected with another worm called Mansonella perstans (Mp). Mp is spread through a biting insect called a midge. It rarely causes symptoms. However, researchers think that Mp infection could affect the body s response to PZQ treatment for or risk of reinfection with Sh.

Objective:

To find out the effects of Mp infection on the response to PZQ treatment for Sh infection.

Eligibility:

Men and women ages 14-80 who:

* Live in Tieneguebougou, Bougoudiana, or surrounding villages in Mali
* Are not pregnant
* Have Sh infection
* Have no other chronic medical conditions

Design:

* Participants will be screened with:

  * Medical history
  * Physical exam
  * Blood and urine tests
  * Stool samples
* Participants will be treated with a single dose of PZQ by mouth.
* After receiving PZQ, participants will return to the clinic for blood and urine tests at the following times:

  * 4, 8, 24, 48, and 72 hours later
  * 5, 7, 9, and 14 days later
  * 1, 3, and 6 months later

Participants who are infected with Sh at the 6-month visit will get another treatment with PZQ.

...

DETAILED DESCRIPTION:
Chronic filarial infection is associated with downregulation of immune responses to both helminth and non-helminth antigens. Praziquantel (PZQ) treatment of schistosomiasis is associated with a dramatic interleukin-5 (IL-5)-dependent increase in eosinophilia that is correlated with resistance to reinfection. We hypothesize that chronic filarial infection with Mansonella perstans (Mp) may attenuate post-treatment eosinophilia and thus impact resistance to reinfection. To address the first part of this question, we plan to compare post-PZQ reactions and reinfection rates in 20 subjects with schistosomiasis and Mp infection to those in 20 subjects with schistosomiasis and no evidence of filarial infection in an area coendemic for both infections in Mali. Signs and symptoms, complete blood counts, intracellular and serum cytokine levels, and markers of eosinophil activation will be assessed at baseline, 4 and 8 hours, and 1, 2, 3, 5, 7, 9, and 14 days post-treatment and compared between the two treatment groups. Schistosoma haematobium reinfection rates will also be compared at 1, 3, and 6 months post-treatment.

ELIGIBILITY:
* INCLUSION CRITERIA (SCREENING):

  1. Male or non-pregnant female subjects
  2. Age 14-80 years (per participant self-report)
  3. Resident of Tienegubougou, Bougoudiana or surrounding villages

  5. Consent to a blood draw to screen for filarial infection and a urine exam to screen for schistosomiasis

  6. Must be willing to have blood samples stored.

EXCLUSION CRITERIA (SCREENING):

1. Known to be pregnant (by history)
2. Chronic medical conditions, including but not limited to diabetes, renal or hepatic insufficiency, immunodeficiency, psychiatric disorder, seizure, that in the investigators judgments are deemed to be clinically significant
3. History of hypersensitivity reaction to PZQ.
4. Weight less than 20 kg

INCLUSION CRITERIA (INTERVENTIONAL STUDY):

1. S. haematobium infection documented at screening and within 14 days prior to the baseline visit
2. The subject agrees to storage of samples for study.

EXCLUSION CRITERIA (INTERVENTIONAL STUDY):

1. Pregnancy (by urine beta-HCG)
2. Chronic kidney or liver disease
3. Hgb <10 mg/dL
4. PZQ treatment since the screening visit
5. Concomitant Schistosoma mansoni, Wuchereria bancrofti (Wb) or Onchocerca volvulus infection
6. Use of immunosuppressive therapies, including steroids, within the past month
7. Any condition that in the investigator s opinion places the subject at undue risk by participating in the study.

EXCLUSION OF CHILDREN AND PREGNANT WOMEN:

Pregnant women will be excluded from this study since it involves administration of medications contraindicated in pregnancy. Children less than 14 years old will be excluded because of the amount of blood required for the immunologic studies. The age of consent in Mali is 18 years of age, so children aged 14 to 17 years will sign an assent form in addition to the consent form to be signed by a parent or tutor. However, married women between the ages of 14 and 17 will sign consent as adults in view of the laws governing emancipation of women in Mali. Subjects who do not participate in this study will receive PZQ as part of the national schistosomiasis control program.

Participation of Women:

-Pregnancy: The effects of praziquantel on the developing human fetus are unknown (pregnancy category B). For this reason, females of

childbearing-age must have a negative pregnancy test result prior to receiving praziquantel. Since the half-life of praziquantel is short (3-4 hours), contraceptive measures will not be required post-treatment.

-Breast feeding: Praziquantel is known to be present in breast milk for up to 3 days following a single dose and is not approved for use in children under the age of 4 years. Consequently, women will be asked to suspend breastfeeding after treatment with PZQ for 3 days. Formula will be provided for breastfed children affected by their mother s participation during this time to ensure adequate nutrition. Depending on the age of the child, formula may be given. A pediatric nurse will be present during this time to provide assistance and counsel to the mothers.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04-06; Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Peak percentage change from baseline eosinophil count | During the first 7 days post-treatment

SECONDARY OUTCOMES:
Peak absolute change from the baseline eosinophil count and peakpercentage change in eosinophil granule protein levels | During the first 7 days post-treatment
Frequency and severity of adverse events | During the first 3 days post-treatment
Number of subjects with detectable Sh eggs in urine | At 1, 3 and 6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)

REFERENCES:
- [Background] Dolo H, Coulibaly YI, Dembele B, Konate S, Coulibaly SY, Doumbia SS, Diallo AA, Soumaoro L, Coulibaly ME, Diakite SA, Guindo A, Fay MP, Metenou S, Nutman TB, Klion AD. Filariasis attenuates anemia and proinflammatory responses associated with clinical malaria: a matched prospective study in children and young adults. PLoS Negl Trop Dis. 2012;6(11):e1890. doi: 10.1371/journal.pntd.0001890. Epub 2012 Nov 1. PMID 23133692
- [Background] Fitzsimmons CM, Joseph S, Jones FM, Reimert CM, Hoffmann KF, Kazibwe F, Kimani G, Mwatha JK, Ouma JH, Tukahebwa EM, Kariuki HC, Vennervald BJ, Kabatereine NB, Dunne DW. Chemotherapy for schistosomiasis in Ugandan fishermen: treatment can cause a rapid increase in interleukin-5 levels in plasma but decreased levels of eosinophilia and worm-specific immunoglobulin E. Infect Immun. 2004 Jul;72(7):4023-30. doi: 10.1128/IAI.72.7.4023-4030.2004. PMID 15213147
- [Background] Keiser PB, Coulibaly YI, Keita F, Traore D, Diallo A, Diallo DA, Semnani RT, Doumbo OK, Traore SF, Klion AD, Nutman TB. Clinical characteristics of post-treatment reactions to ivermectin/albendazole for Wuchereria bancrofti in a region co-endemic for Mansonella perstans. Am J Trop Med Hyg. 2003 Sep;69(3):331-5. PMID 14628953